CLINICAL TRIAL: NCT00351676
Title: Capturing Outcomes of Clinical Activities Performed by a Rounding Pharmacist Practising in a Team Environment (COLLABORATE)
Brief Title: Capturing Outcomes of Clinical Activities Performed by a Rounding Pharmacist Practising in a Team Environment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Capital Health, Canada (Other)
Responsible Party: Dr. Ross Tsuyuki, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: EPICORE-2006-001
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2006-02

CONDITIONS: Heart Failure, Congestive; Pulmonary Disease, Chronic Obstructive; Pneumonia; Diabetes Mellitus, Type 2; Coronary Arteriosclerosis
Keywords: Drug Therapy; Hospitals, Teaching; Hospitals, Community; Interprofessional relations; Patient Care Team; Pharmacists; Pharmacy Service, Hospital; Comparative Study; Hospitalization
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Pneumonia; Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Integration of a team based clinical pharmacist
Drug: Optimizing therapeutic treatments
Behavioral: Optimizing processes of care

SUMMARY:
We, the researchers, propose to link a clinical pharmacist with an internal medicine or family medicine team to provide pharmaceutical care to all patients assigned to the team. The hypothesis is that through this team based approach, pharmacists will act as a resource for providing pharmacotherapeutic advice during the drug therapy decision making process and promote optimal drug use by identifying and resolving actual and potential drug related problems. This study is designed to test this hypothesis, by assessing the impact of this intervention on evidence based, quality of drug therapy indicators, for patients admitted with heart failure (HF), chronic obstructive pulmonary disease (COPD), community acquired pneumonia (CAP), type 2 diabetes mellitus (T2DM), and stable coronary artery disease (CAD).

DETAILED DESCRIPTION:
The overall goal of the COLLABORATE study is to improve processes of care and patient outcomes by optimizing drug therapy via a hospital pharmacy practice model that integrates clinical pharmacists into the patient care team.

The intervention consists of a clinical pharmacist assigned to the patient care team for the purpose of providing proactive clinical pharmacy services. The study pharmacist will be available during normal office hours 5 days per week to provide clarification of the patient's medication history, identify and resolve actual and potential patient specific drug related problems/issues, participate in patient care rounds, provide drug information to the patient care team, provide patient education and discharge medication counselling, and provide physician and/or nursing staff education. The anticipated pharmacist to patient ratio is approximately 1:20.

Control patients will receive usual care. Usual care consists of reactive clinical pharmacy services (i.e. drug related issues identified as orders are received, or by patient profile review) provided by a ward based, not team based, clinical pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients > 18 years of age admitted to participating internal and family medicine teams during the 1 year study period will be eligible to receive the pharmacist intervention. For the purposes of data analysis, patients with a most responsible or primary diagnosis of HF, COPD, CAP, T2DM, and CAD will be included.

Exclusion Criteria:

* Residence outside the Capital Health catchment
* Admitted for ≤ 2 days
* Palliative care
* Transferred to another team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2006-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Improvement in proportion of quality indicators achieved, for target diseases as a most responsible or primary diagnosis, between groups. | in hospital

SECONDARY OUTCOMES:
Differences in condition-specific achievement of drug therapy quality indicators; | in hospital
Differences in 6 month hospital readmission rate; | 6 months
Differences in number, type, acceptance rate, and expected impact of all pharmacist interventions; | in hospital
Qualitative evaluation of the impact of the intervention via interviews with the participating pharmacists and physicians. | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ross T. Tsuyuki, PharmD, MSc, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta

REFERENCES:
- [Derived] Makowsky MJ, Koshman SL, Midodzi WK, Tsuyuki RT. Capturing outcomes of clinical activities performed by a rounding pharmacist practicing in a team environment: the COLLABORATE study [NCT00351676]. Med Care. 2009 Jun;47(6):642-50. doi: 10.1097/MLR.0b013e3181926032. PMID 19433997
- [Derived] Makowsky MJ, Schindel TJ, Rosenthal M, Campbell K, Tsuyuki RT, Madill HM. Collaboration between pharmacists, physicians and nurse practitioners: a qualitative investigation of working relationships in the inpatient medical setting. J Interprof Care. 2009 Mar;23(2):169-84. doi: 10.1080/13561820802602552. PMID 19234987
- See also: Related Info — https://www.epicore.ualberta.ca